CLINICAL TRIAL: NCT01655875
Title: A Pilot Study of AMD3100 as a Sensitizing Agent in Myeloablative Allogeneic Blood and Marrow Transplantation for Chemotherapy Resistant Pediatric Acute Leukemia
Brief Title: AMD3100 for Sensitizing in Allogeneic Blood or Marrow Transplant for Chemotherapy Resistant Pediatric Acute Leukemia
Acronym: BMTAMD3100
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of patient enrollment
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kuang-Yueh Chiang, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00053638; CHOA AMD3100 Pilot (Other: Other)
Record Dates: First submitted 2012-07-27; First posted 2012-08-02 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Pediatric Acute Myeloblastic Leukemia, Relapsed; Pediatric Acute Lymphoblastic Leukemia, Relapsed
Keywords: Allogeneic Blood and Marrow Transplantation
MeSH Terms: conditions — Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bone marrow transplant (Experimental)
  Interventions: Drug: AMD3100

INTERVENTIONS:
Drug: AMD3100 — AMD3100 will first be administered at 240 mcg/kg (the FDA approved dose for mobilization of autologous PBSC) IV once daily prior to conditioning for 3 days (days -6, -5 and -4) in the first group of participants. If toxicity criteria are met, the dosing will be escalated in the second group of participants to 240 mcg/kg IV once daily prior to conditioning for 5 days (days -8, -7, -6, -5 and -4).
  Other Names: Mozobil; Plerixafor

SUMMARY:
This study is for patients 2-21 years old who have acute leukemia that has not responded well to chemotherapy and will have a bone marrow transplant. This is a pilot (phase 1) study of AMD3100(also called Plerixafor, Mozobil). AMD3100 is given in combination with a standard pre-transplant conditioning regimen (total body irradiation, etoposide and cyclophosphamide). The conditioning regimen is the treatment that is given just before the transplant. This treatment kills leukemia cells as well as healthy bone marrow and immune cells. Researchers want to learn more about how AMD3100 affects acute leukemia cells. Blood and bone marrow samples from study participants will be collected to find out if AMD3100 is making patients' cells more sensitive to the conditioning regimen and to find out how it does this.

The first six patients receive three daily doses (240 mcg/kg via IV). If it appears that three doses do not significantly increase the side effects of transplant conditioning, the investigators will give a second group of six patients five daily doses.

DETAILED DESCRIPTION:
The first six patients will receive three daily doses of AMD3100 (240 mcg/kg via IV). If it appears that three doses do not significantly increase the side effects of transplant conditioning, the investigators will give a second group of six patients five daily doses.

AMD3100 is given in combination with a standard pre-transplant conditioning regimen (total body irradiation, etoposide and cyclophosphamide.) AMD3100 causes healthy bone marrow cells to be released from the bone marrow into the blood so that they can be collected in patients who will have peripheral (blood stream) blood stem cell transplants. AMD3100 also pushes out leukemia cells from the bone marrow. Research in animals and in test tubes shows that the bone marrow partially protects leukemia cells from chemotherapy and radiation. AMD3100 could make leukemia treatments better by pushing out the leukemia cells from the bone marrow and making them more sensitive to treatment. Clinical trials combining AMD3100 with normal doses of chemotherapy are being done for relapsed acute leukemia. Researchers hope AMD3100 can be given with conditioning regimen safely without causing more side effects. Up to 12 participants will be enrolled and estimated accrual duration is 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Must have chemotherapy-resistant acute leukemia (primary refractory or relapsed and refractory AML, ALL, undifferentiated, bi-lineage or mixed lineage leukemia)
* Participant must have a well HLA matched related, mismatched related or unrelated marrow donor with whom the patient is allele matched at at least 7 of 8 HLA loci or a single unrelated cord blood unit matched at at least 4 of 6 HLA loci with minimal dose of 4x10(7)NC/Kg

Exclusion Criteria:

* Prior allogeneic or autologous hematopoietic stem cell transplantation
* Prior exposure to AMD3100
* Active central nervous system leukemia
* Uncontrolled viral, bacterial, fungal, protozoal infection
* HIV infection
* Does not meet standard organ function for transplant

Ages: 2 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
AMD3100 safety | day 42 after bone marrow transplant
  Incidence of grade 3 and 4 regimen-related toxicity assessed per Bearman scale at day 42. Patients in dose level 1 get 3 days of AMD3100. If 2 cases of grade 4 toxicity or 3 cases of grade 3-4 toxicity occur, dose level 1 and study will be closed. Otherwise, after 6 patients have been assessed at day 42, the dose will be escalated to 5 days of AMD3100 (dose level 2). If 2 cases of grade 4 toxicity or 3 cases of grade 3-4 toxicity occur, the study will be closed. Otherwise, after 6 patients have been enrolled at this level the study will be closed to enrollment.

SECONDARY OUTCOMES:
AMD3100 correlative biology analyses | 2 years
  Bone marrow and peripheral blood samples collected during study are examined in the laboratory to detect if there is any difference in leukemia cells after treatment with AMD3100.

CONTACTS AND LOCATIONS:
Overall Officials: Kuang-Yueh Chiang, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States